CLINICAL TRIAL: NCT00452894
Title: A Pharmacokinetic, Toleration And Safety Study Of Single And Multiple Oral Doses Of Varenicline In Chinese Healthy Volunteers
Brief Title: Phase 1 Clinical Trial of Varenicline in Chinese Healthy Smoking Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3051076
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline tartrate

SUMMARY:
This study is to measure how much of varenicline tartrate is in Chinese healthy smokers' blood and urine after taking a single dose and several doses respectively, and also to test the safety (the impact of the study drug on Chinese healthy smokers' body) of varenicline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female Chinese subjects between the ages of 18 and 45 years, inclusive.
* Body Mass Index (BMI) of approximately 19 to 24 kg/m2; and a total body weight ≥50 kg.
* Individuals who have smoked an average of at least 10 cigarettes per day during the past year, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Heart rate>100 bpm, QRS Interval>120 msec, QTc Interval >430 msec, PR Interval>220 msec, or any other abnormalities observed on the Electrocardiogram.
* Subjects with a sitting blood pressure of 140/90 mmHg or above at screening.
* Subjects with evidence or history of clinically significant allergic, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric or neurological disease, or any condition possibly affecting drug absorption.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14
Dates: Start 2007-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The PK parameters after a single dose and PK parameters after 7 days of multiple dosing respectively.

SECONDARY OUTCOMES:
To gather safety data from Day 0 to Day 17 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Beijing, China

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051076&StudyName=Phase+1+Clinical+Trial+of+Varenicline+in+Chinese+Healthy+Smoking+Volunteers+